CLINICAL TRIAL: NCT04253782
Title: A Multi-Tiered Safety Net Following Naloxone Resuscitation From Opioid Overdose
Brief Title: SafetyNet Program for Opioid Use Disorder (OUD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000028548; R01CE002989-01 (NIH); 2000027149 (Other: OTHER YALE IRB IDENTIFIER)
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Opioid-Use Disorder (OUD)
Keywords: Community Healthcare; Emergency Medicine; Addiction Recovery; Substance Misuse; Opioid Overdose
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose

STUDY DESIGN:
Intervention Model Description: Study personnel (recovery coaches + health educators) will form teams and meet (mostly remotely/electronically and/or by phone) with participants, who will select one of three options that may help with opioid misuse:
  1. treatment with buprenorphine/naloxone (BUP),
  2. methadone maintenance, intensive outpatient, or residential treatments, or
  3. education only. Throughout the study, participants may switch to any other option.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Team Intervention Arm (Experimental): Recovery coaches and trained health educators will team together and meet with participants (remotely/electronically and/or by phone or in person, when appropriate) at least twice and for a maximum of 7 times. This includes access to mediation, trained mental healthcare providers, and educational resources.
  Interventions: Other: Team Intervention

INTERVENTIONS:
Other: Team Intervention — The Team will meet with participants (remotely/electronically and/or by phone) and will ask that they select one of three options that may help with opioid addiction:
  1. treatment with buprenorphine/naloxone (BUP),
  2. inpatient, 12-step, or methadone regimens, or
  3. education only (materials provided by the CT Community for Addiction Recovery (CCAR)).
  Throughout the study, participants may switch to any other option.

SUMMARY:
The principal aim of this study is to determine whether a novel biopsychosocial intervention following opioid overdose (OD) affects 1) the frequency of secondary opioid OD events and 2) the proportion of individuals who remain engaged in treatment for opioid use disorder (OUD) or are in remission at 30 days and at 180 days post intervention. Remission is defined as engagement in daily medication-assisted therapy (MAT)-typically buprenorphine/naloxone (BUP) or methadone- and/or a recovery capital score of ≥ 27.5. The intervention principally involves connecting OUD-affected individuals with community resources, including BUP-, other MAT-, and education-related services. To carry out the intervention, an addiction recovery coach and an appropriately trained health educator paramedic (research assistant) will form a Team and perform follow-up visits (electronically/remotely and/or by phone and/or in person, when appropriate) after a participant has experienced at least 1 opioid OD requiring naloxone resuscitation. Our hypothesis is that the intervention will decrease subsequent OD events and increase the likelihood of remission. To evaluate this hypothesis, data will be collected from self-report and from EPIC, Yale New Haven Hospital's medical record system. The secondary aim is to determine whether the intervention affects 1) the frequency of positive-urine tests for opioids and 2) the frequency and proportion of subjects self-reporting opioid use. Our hypothesis is that this intervention will decrease both. Data from the entire cohort will be compared in aggregate with patients who were started on BUP in the ED over the same time period and with historic controls.

DETAILED DESCRIPTION:
Scientific premise for proposed project. Buprenorphine/naloxone-based (BUP) treatment for opioid use disorder (OUD). It is known that medication-assisted therapy (MAT) of opioid use disorder (OUD) with buprenorphine/naloxone (BUP) is associated with decreased risk of opioid overdose, improved engagement in treatment at 30 days, and less self-reported opioid use compared with those who receive only a brief negotiated interview (BNI) or referral for counselling. As a result of previous research, patients in Yale's Emergency Department (ED) who are successfully resuscitated with naloxone following an opioid overdose are routinely screened using the Mini International Neuropsychiatric Interview (MINI) for OUD. Those who screen positive for moderate to severe OUD are offered initiation of BUP treatment in the ED, with outpatient primary care clinic referral for ongoing medical monitoring and treatment. At the time of the ED visit, however, fewer than half of these patients will consent to initiation of BUP. Those who decline are offered overdose education and naloxone (OEN) by ED staff. A safety net that includes tailored linkage plans to effectively engage opioid overdose survivors with BUP, intensive psychosocial support, and follow-up counseling in the community is needed. To gain a better understanding of the motivations of those who decline the offer of BUP, research from Yale's Department of Emergency Medicine purposively sampled 16 opioid overdose survivors who agreed to participate in a qualitative study looking at their knowledge and understanding of OUD (unpublished). Predominant themes included the following: ambivalence regarding the effectiveness of treatment for OUD, concerns about concurrent social supports such as housing and mental health services; lack of appreciation for the risks associated with OUD (even with multiple prior overdoses); strong, but abstract, desire to discontinue use of opioids, despite refusal of treatment; and limited understanding of how to prevent or emergently manage overdoses. These perceptions from the patient population with OUD declining treatment directly informed the current study and its proposed research strategy.

Peer support and recovery in OUD. In 2012, the Substance Abuse and Mental Health Services Administration (SAMHSA) established a working definition of recovery from mental health and substance use disorders: a process of change through which individuals improve their health and wellness, live self-directed lives, and strive to reach their full potential. The definition identifies 4 dimensions that support recovery: 1) health, including both management of the disease and decision making associated with physical and emotional wellbeing; 2) home, e.g., a stable place to live; 3) purpose, e.g., meaningful daily activities; and 4) community, e.g., supportive relationships and social networks. One of the interrelated guiding principles of recovery promulgated by SAMHSA is peer support. Peer recovery support services are delivered by persons who have common life experiences with those they are serving. Since 1998, SAMHSA has sponsored Recovery Community Services grant programs, and in 2002 the program changed its focus to emphasize the use of peers for recovery support services. This funding now targets recovery community statewide networks. The Connecticut Community for Addiction Recovery (CCAR) was established in 1998, with initial funding by the State's Department of Mental Health and Addiction Services and one of the original SAMHSA grants. Since then, it has grown to its current size with a staff of 28, recovery centers located in major cities, an ED recovery coach program, and 308 volunteers who donated 28,841 hours in 2017 alone. CCAR recovery coaches are peer experts; many have been in recovery themselves. They have experiential knowledge and training. More specifically, CCAR describes a recovery coach as a motivator who exhibits bold faith in an/a individual/family's capacity for change, and who encourages and celebrates achievement. The recovery coach is an ally and confidant who genuinely cares, listens, and can be trusted with confidences, as well as a truth teller who provides a consistent source of honest feedback regarding self-destructive patterns of thinking, feeling, and acting. He or she is also a role model and mentor who offers his/her life as living proof of the transformative power of recovery and provides stage-appropriate recovery education and advice. The recovery coach is trained to serve as a problem solver who identifies and helps remove personal and environmental obstacles to recovery. He or she serves as a resource broker, linking individuals/families to formal and indigenous resources such as sober housing, recovery-conducive employment, health and social services, and other recovery support. The recovery coach advocates by helping individuals and families navigate service systems for access, responsiveness, and protection of rights. The recovery coaches may also be community organizers to help develop and expand available recovery support resources, lifestyle consultants to assist individuals/families to develop sobriety-based rituals of daily living, and friends, providing companionship. Coaches receive training at the CCAR Recovery Coach Academy, a 5-day intensive training program that focuses on providing individuals with the necessary skills to mentor, support, and guide any person who would like to enter or sustain long-term recovery from addiction. At this training, prospective CCAR recovery coaches learn about the roles and functions of a recovery coach, core values and guiding principles of recovery, relationship enhancement and crafting skills, appropriate attitudes about self-disclosure, stages of recovery, addressing stigma, awareness of culture, power and privilege, and addressing ethical and boundary issues. This Academy also teaches how to practice newly acquired skills. CCAR recovery coaches' style of treatment is generally informal, and they assist the individual affected by OUD in focusing on what he or she can do at the present time to facilitate recovery in the future, in addition to helping these individuals connect with community resources. Reports suggest that fostering a supportive and positive treatment environment is critical.

Community treatment of OUD. Some small studies and anecdotal successes have been reported in a variety of settings when community health educators were included in programs to assist patients with OUD. Most of the available reports are in emergency medical services (EMS) trade journals, organization newsletters, public news releases, and other "gray" literature. For example, a Fairfield County, Ohio initiative called Project FORT (Fairfield Overdose Response Team) dispatches a community paramedic and a law enforcement officer to meet with patients after opioid overdoses. This is a community outreach model program that contacts patients, within 1-3 days of overdose, and assists them with getting into treatment facilities, which are aimed primarily at abstinence. With no reports of formal outcomes, as of December, 2017, Project FORT had piloted 12 patients. Of these, 1 was known to be in an inpatient treatment program, and another had been admitted to the hospital for opioid withdrawal then discharged to inpatient treatment. The Johns Hopkins Bloomberg School of Public Health is collaborating with Baltimore City Fire Department's paramedics and the Behavioral Health System of Baltimore in a program that trains the paramedics to perform a screening test for OUD, followed by a BNI after responding to opioid overdoses. At the time of their report, patients with OUD were being referred by the paramedics to a community-based research center within the Bloomberg School for counseling, motivation, and discussion of barriers to treatment. HIV (+) patients were preferentially referred to a medical facility for treatment with BUP along with management of their HIV disease. Their longer-term plan was to eventually transport clinically stable patients after overdose directly to a sobering center, similar to the protocol used in the City of San Francisco. Although the patients referred by the paramedics to the community-based research center are randomized to one of 2 different treatment arms, there have been no reports of the effectiveness of the paramedics in this role. In a Palm Beach, FL community paramedicine program loosely based on previous work at Yale, consented patients are started on BUP in the ED after an overdose. But community paramedics deliver the ensuing daily doses to the patients at home for the first week of therapy. These medics are accompanied by peer recovery specialists who work with the patient on support systems for longer term recovery. Although no outcomes data are available for this program, it involves a rapid taper off of BUP early in the treatment regimen. In most other studies, early discontinuation of BUP is associated with poorer short- and long-term outcomes, and increased risk of nonfatal and fatal overdoses.

The Paramedic Referrals for Increased Independence and Decreased Disability in the Elderly (PRIDE) program at Yale. Findings from the Department of Emergency Medicine previously demonstrated that 1/3 of all seniors who activated the local 9-1-1 system due to inability to get up after a fall at home would activate 9-1-1 again within the ensuing 30 days. Furthermore, 2/3 of all calls to EMS for a "lift assist" were repeat calls to the same address within the previous 30 days. By addressing some of the factors contributing to the risk of falling, and by improving access to community medical resources based on individuals' needs, many unplanned healthcare encounters likely could be prevented, while keeping participants safely in their homes. Thus, a collaborative program between research paramedics and home healthcare nurses was established. The program was funded by a Health Care Innovations Award from the Centers for Medicare & Medicaid Services in 2014. The overarching goal of Paramedic Referrals for Increased Independence and Decreased Disability in the Elderly (PRIDE) was to help older individuals to live independently, while decreasing requirements for unplanned utilization of EMS, EDs, and hospitalization. To be eligible to participate in PRIDE, seniors must have fallen in the past or felt that they were at risk for falling, resided within a 15-town area in South-Central Connecticut, and resided at home or in an assisted-living facility. The program's intervention involved home visits by the PRIDE Team. Health-educator paramedics, as research assistants, and nurses recorded results of balance and other agility tests, participants' medications, vital signs, and performed safety assessments of the living space. The home healthcare nurses evaluated gait, posture, cardiovascular health and medications, requirements for durable medical equipment, and ongoing care needs, such as physical or occupational therapy. All participant data were entered into a Health Insurance Portability and Accountability (HIPAA)-compliant, encrypted database: Research Electronic Data Capture (REDCap). Additionally, if needed, staff set up appointments with the participant's primary care provider, and a free ride in a medically appropriate vehicle to and from the appointment was included. Subsequent unplanned healthcare utilization was tracked using the electronic medical record system at Yale New Haven Hospital (YNHH). PRIDE operated from 2014-2018 and enrolled greater than 5,600 participants. Data (currently unpublished) to date demonstrate that there are significantly fewer ED visits and less EMS utilization among those who received PRIDE services, compared with participants who enrolled but declined visits by PRIDE staff. These data suggest that PRIDE's intervention was effective in decreasing unplanned healthcare utilization.

Proposed adaptation of PRIDE to serve persons with OUD. We propose to adapt the PRIDE program infrastructure to provide a safety net for patients who 1) have been resuscitated from an opioid overdose with naloxone, 2) have screened positive for OUD using the MINI, and 3) refused to initiate treatment with BUP in the ED, if offered. We may also include and accept referrals from CCAR, Project Alcohol & Substance Abuse Services, Education, and Referral to Treatment (ASSERT) (whose recruiters work in the YNHH EDs), staff working in the Yale EDs and with American Medical Response (AMR) units, and a Community Health Care Van. For this program, the composition of the field teams will be changed, pairing recovery coaches from CCAR with experienced PRIDE research paramedics, to form RCP Teams. For those affected by moderate-severe OUD, we expect that engaging with the RCP Teams will create a more robust linkage of care with community resources and treatment options. Importantly, these Teams will motivate interest in treatment, facilitate access to BUP or methadone or equivalent, assist with other community-based recovery strategies, help address acute psychosocial issues, and provide ongoing education and counselling. The requirements for these capabilities were derived from our previous qualitative studies of persons with OUD who declined ED-initiated treatment.

Research plan. To date, there is no standard of care for individuals with OUD who have overdosed on opioids, have been resuscitated by naloxone, and have refused BUP treatment. As noted previously, YNHH typically will send home these individuals with OEN kits. However, follow-up care remains variable. Hence, this research seeks to determine whether individuals with OUD might benefit significantly from a novel, Team-based intervention encouraging biopsychosocial and medical interventions. First, this work will assess whether a novel biopsychosocial intervention following OD affects 1) the frequency of secondary opioid OD events and 2) the proportion of individuals who remain engaged in treatment for OUD or are in remission within 30 and 180 days post intervention. Remission may be defined as engagement in daily medication-assisted therapy-typically buprenorphine/naloxone (BUP) or methadone- and/or a recovery capital score of ≥ 27.5. The study's hypothesis is that the intervention by the RCP team will decrease subsequent OD events and increase the likelihood of remission. This work also seeks to determine whether the intervention affects 1) the frequency of positive-urine tests for opioids and 2) the frequency and proportion of subjects self-reporting opioid use. The hypothesis is that the intervention will decrease both. The study plan is as follows: To prepare for the intervention, health educators and key study staff are required to attend 12 hours of in-person training, which is to take place over 2 days, to learn about best practices assessing those with OUD. One of the co-principal investigators (co-PIs) of this study, along with CCAR staff, will teach. Sessions will include training to conduct a BNI and a brief assessment of recovery capital (BARC-10) interview. Training also will prepare all staff to respectfully ask questions about potential overdose events and the possibility of creating and/or implementing a wellness plan. After resuscitation from opioid overdose by naloxone individuals in the EDs at the York St. and Chapel St. campuses of YNHH will be screened by ED providers for OUD using a MINI. This is an evidence-supported, standard practice at Yale. Upon screening positive for OUD, individuals should be offered BUP treatment by staff. Those who screen positive for OUD, but who decline BUP, will be offered overdose and naloxone kits. In addition, the study Team will approach these individuals to ask whether they might be interested in research participation. If the patient were to express interest, then the study Team members would set up an appointment (remotely/electronically and/or by phone and/or in person, if appropriate) to meet at a time and place of the prospective/ participant's choosing. Depending on preference informed consent may be obtained in the ED or at the first outpatient visit. In addition, individuals from CCAR may refer interested individuals to study participation, providing that at some time in the previous 7 days they had overdosed on opioids, were resuscitated by naloxone, and screened positive for OUD in a YNHH ED. After consent and study initiation, either at the hospital or later, the Team will perform a BNI- whose goal is to employ motivational techniques to help those with substance misuse consider their reasons for wanting to address dependency. The Team will perform psychosocial and medical evaluations. The Team will also enter all data into a secured, encrypted database, REDCap. Approximately 30 days after consent, the Team will schedule Meeting 1 with participants. During this time, the Team will collect and enter data into REDCap based on discussions with and evaluations of participants. During Meeting 2, which should occur no more than 180 days after consent, the Team will also collect and enter data into REDCap based on discussions with and evaluations of participants. The study team will also enter data from participants' medical records at all time intervals. Because of the COVID-19 outbreak, at the time of this writing (07/25/2020), many follow-up visits will occur remotely/electronically, using HIPAA-compliant software + data bases, and/or by phone. However, on a case-by-case basis, in-person follow up visits are permitted.

Data from the entire cohort will be compared in aggregate with patients who were started on BUP in the ED over the same time period and with historic controls.

COVID-19 restrictions and other logistical challenges impacted the completion of the study; including the ability to collect and report the outcome measures as intended in the original proposed research. In part, patient self-report outcomes were not collected. In addition, upon the entry of results at study termination, the outcomes were updated to reflect those that were omitted in the original protocol registration. All of the outcomes reported reflect the information that could be obtained from the Electronic Health Record given the interruption of study procedures.

Due to limitations that arose during the study, many of which were related to the COVID pandemic which unfortunately broke out just as the study was preparing to launch, this study had to be significantly modified. Investigators performed a prospective study following the individuals who accepted the intervention. Historical controls were used only to calculate a desired sample size, but were not used to compare outcomes. Investigators did not compare directly to individuals enrolled in BUP during the same period. This study was simply presented this as a possible alternative approach and results were entered.

ELIGIBILITY:
Inclusion criteria

1. ≥18 years
2. Screen positive for opioid use disorder (OUD)
3. Screen positive for OUD using the mini international neuropsychiatric interview (MINI)
4. At least 1 opioid overdose requiring resuscitation by naloxone or equivalent
5. No non-opioid overdose explanation for decreased level of consciousness, miosis, or decreased respiratory rate
6. Positive for OUD using a health questionnaire containing questions about prescription opioid and heroin use
7. Not in a critically ill state at the time of consent (e.g., not actively suicidal, psychotic, septic, nor cardiac arrest; nor any combination; nor equivalent)
8. 3., 4., & 6. (in III. Inclusion criteria) must have occurred within ≤7 days (inclusive) from the date of consent if the prospective participant were discharged from the hospital or equivalent treatment facility
9. Not homicidal
10. Able to self-consent to program/study participation
11. Permanent residence is not a long-term care facility
12. No simultaneous enrollment in another study whose principal investigator (PI) or co-PI is a faculty member in the Department of Emergency Medicine at the Yale School of Medicine
13. Not prescribed opioids for acute pain, chronic pain, or palliative care without OUD diagnosis
14. Not stably enrolled in opioid agonist treatment for OUD at the time of the ED visit
15. Neither in police custody nor incarcerated nor both; nor equivalent; *parolees and those on probation may be enrolled incidentally, but are not the target population of this work
16. Refused buprenorphine/naloxone (BUP), if offered
17. Has a valid mailing address or P.O. box
18. Able to answer questions electronically/remotely, by phone, or by any combination of these technologies

Exclusion criteria

1. <18 years
2. Screen negative for OUD
3. Screen negative for OUD using the mini international neuropsychiatric interview (MINI)
4. No evidence of documented opioid overdose requiring resuscitation by naloxone or equivalent
5. Non-opioid overdose explanation for decreased level of consciousness, miosis, or decreased respiratory rate
6. Negative for OUD using a health questionnaire containing questions about prescription opioid and heroin use
7. In a critically ill state (e.g., actively suicidal, psychotic, septic, or in cardiac arrest; any combination; or equivalent) at the time of consent
8. 3., 4., & 6. (in III. Inclusion criteria) have occurred >7 days (exclusive) from the date of consent if the prospective participant were discharged from the hospital or equivalent treatment facility
9. Homicidal
10. Unable to self-consent to program/study participation
11. Permanent resident of a long-term care facility
12. Simultaneous enrollment in another study whose principal investigator (PI) or co-PI is a faculty member in the Department of Emergency Medicine
13. Prescribed opioids for acute pain, chronic pain, or palliative care without OUD
14. Stably enrolled in opioid agonist treatment or other medication-assisted therapy for OUD at the time of consent
15. In police custody and/or incarcerated or equivalent; *parolees and those on probation may be enrolled incidentally, but are not the target population of this work
16. On BUP treatment
17. No valid mailing address or P.O. box
18. Unable to answer questions electronically/remotely, by phone, or by any combination of these technologies

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Joseph, MD, Principal Investigator — Yale University School of Medicine, Yale New Haven Hospital
Locations (2):
- United States (2):
  - Yale New Haven Hospital, 20 York Street, New Haven, Connecticut
  - Yale New Haven Hospital, Saint Raphael Campus, 1450 Chapel Street, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Onofrio G, O'Connor PG, Pantalon MV, Chawarski MC, Busch SH, Owens PH, Bernstein SL, Fiellin DA. Emergency department-initiated buprenorphine/naloxone treatment for opioid dependence: a randomized clinical trial. JAMA. 2015 Apr 28;313(16):1636-44. doi: 10.1001/jama.2015.3474. PMID 25919527
- [Background] Dugosh K, Abraham A, Seymour B, McLoyd K, Chalk M, Festinger D. A Systematic Review on the Use of Psychosocial Interventions in Conjunction With Medications for the Treatment of Opioid Addiction. J Addict Med. 2016 Mar-Apr;10(2):93-103. doi: 10.1097/ADM.0000000000000193. PMID 26808307
- [Background] Amorim P, Lecrubier Y, Weiller E, Hergueta T, Sheehan D. DSM-IH-R Psychotic Disorders: procedural validity of the Mini International Neuropsychiatric Interview (MINI). Concordance and causes for discordance with the CIDI. Eur Psychiatry. 1998;13(1):26-34. doi: 10.1016/S0924-9338(97)86748-X. PMID 19698595
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Substance Abuse and Mental Health Services Administration. SAMHSA's working definition of recovery: 10 guiding principles of recovery. 2012. PEP12-RECDEF https://store.samhsa.gov/system/files/pep12-recdef.pdf (Accessed 1/27/2020)
- [Background] Substance Abuse and Mental Health Services Administration (SAMHSA). What are peer recovery support services? US Department of Health and Human Services; HHS Publication SMA 09-4454. http://www.samhsa.gov/recovery/peer-support-social-inclusion (Accessed 01/27/2020)
- [Background] Kaplan l, Nugent C, Baker M, Clark HW, Veysey BM. Introduction: The recovery community services program. Alcoholism Treatment Quarterly 28: 244-255, 2010.
- [Background] CONNECTICUT COMMUNITY FOR ADDICTION RECOVERY (CCAR). What is a recovery coach? https://addictionrecoverytraining.org/recovery-coach-academy/ (Accessed 01/27/2020)
- [Background] CONNECTICUT COMMUNITY FOR ADDICTION RECOVERY (CCAR). Recovery Coach Academy © https://addictionrecoverytraining.org/recovery-coach-academy/ (Accessed 01/27/2020)
- [Background] Capozzi J. Heroin epidemic: As deaths rise, program a 'glimmer of hope' for life. myPalmBeachPost. https://www.palmbeachpost.com/news/heroin-epidemic-deaths-rise-program-glimmer-hope-for-life/c8ITU5Q2lJbVFfEjSZKwpK/ (Accessed 01/27/2020)
- [Background] Tracy K, Wallace SP. Benefits of peer support groups in the treatment of addiction. Subst Abuse Rehabil. 2016 Sep 29;7:143-154. doi: 10.2147/SAR.S81535. eCollection 2016. PMID 27729825
- [Background] Hayes M. Fairfield County program targets opioid addiction. This Week Community News; Dec 12, 2017. http://www.thisweeknews.com/news/20171212/fairfield-county-program-targets-opioid-addiction (Accessed 01/27/2020)
- [Background] Rienzi G. Johns Hopkins pilots study on EMS treatment of substance abusers. Johns Hopkins University Gazette. Sept-Oct 2014. https://hub.jhu.edu/gazette/2014/september-october/focus-baltimore-city-ems/ (Accessed 01/27/2020)
- [Background] Cone DC, Ahern J, Lee CH, Baker D, Murphy T, Bogucki S. A descriptive study of the "lift-assist" call. Prehosp Emerg Care. 2013 Jan-Mar;17(1):51-6. doi: 10.3109/10903127.2012.717168. Epub 2012 Sep 12. PMID 22971148
- [Background] Yale University Section of EMS. Yale PRIDE. http://www.pride-ems.org/myself/ (Accessed 01/27/2020)
- [Background] Boscarino JA, Kirchner HL, Pitcavage JM, Nadipelli VR, Ronquest NA, Fitzpatrick MH, Han JJ. Factors associated with opioid overdose: a 10-year retrospective study of patients in a large integrated health care system. Subst Abuse Rehabil. 2016 Sep 16;7:131-141. doi: 10.2147/SAR.S108302. eCollection 2016. PMID 27695382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to COVID interruptions investigators only looked at the total number of patients that enrolled in the study which was 81, then compared differences between those who were successfully followed up and those who were not. (This was only among individuals who enrolled in the study.) There were no comparisons made to historic controls or to patients who accepted BUP in the ED during that time period.
Groups:
- SafetyNet Without Successful Follow Ups: Participants that received SafetyNet and had unsuccessful follow-ups.
- SafetyNet With Successful Follow Ups: Participants that received SafetyNet and had successful follow-ups.
Period: Overall Study
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Started | 36 | 45
Completed | 34 | 45
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups | Total
Number analyzed (Participants) | 36 | 45 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.50 (10.49) | 41.62 (11.15) | 39.79 (10.99)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 21 | 34 | 55
  Gender: Female | 14 | 11 | 25
  Gender: Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 10 | 10 | 20
  Race/Ethnicity: White | 20 | 23 | 43
  Race/Ethnicity: Hispanic | 6 | 11 | 17
  Race/Ethnicity: Other/Unlisted | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 45 | 81
Insurance [Count of Participants; unit: Participants]
  Private | 3 | 4 | 7
  Medicare | 2 | 4 | 6
  Medicaid | 30 | 36 | 66
  None | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Positive Urine Tests at 30 Days (Chart Review)
Description: Count of positive urine tests at 30 days after intervention per patient (data obtained via chart review)
Time Frame: 30 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants
  0 positive tests | 35 | 45
  3 positive tests | 1 | 0

2. Primary Outcome: Frequency of Positive Urine Tests at 180 Days (Chart Review)
Description: Count of positive urine tests at 180 days after intervention per patient (data obtained via chart review)
Time Frame: 180 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants
  0 positive tests | 31 | 42
  1 positive test | 2 | 3
  2 positive tests | 1 | 0
  3 positive tests | 1 | 0
  4 positive tests | 1 | 0

3. Primary Outcome: Frequency of Emergency Department Overdose(s) at 30 Days (Chart Review)
Description: Count of Emergency Department Overdose(s) at 30 days after intervention per patient (data obtained via chart review)
Time Frame: 30 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants
  0 overdoses | 32 | 39
  1 overdose | 2 | 3
  2 overdoses | 2 | 2
  3 overdoses | 0 | 1

4. Primary Outcome: Frequency of Emergency Department Overdose(s) at 180 Days (Chart Review)
Description: Count of Emergency Department Overdose(s) at 180 days after intervention per patient (data obtained via chart review)
Time Frame: 180 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants
  0 overdoses | 27 | 34
  1 overdose | 5 | 4
  2 overdoses | 0 | 4
  3 overdoses | 2 | 1
  4 overdoses | 1 | 0
  5 overdoses | 1 | 0
  6 overdoses | 0 | 1
  9 overdoses | 0 | 1

5. Primary Outcome: Percentage of Patients Engaged in Medication Assisted Therapy (MAT) Within 180 Days (Chart Review)
Description: Percentage of patients engaged in Medication Assisted Therapy (MAT) within 180 days after intervention (data obtained via chart review)
Time Frame: 180 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants | 23 | 32

6. Primary Outcome: Percentage of Patients With Any Use of Suboxone Within 180 Days (Chart Review)
Description: Percentage of patients with any use of Suboxone within 180 days after intervention (data obtained via chart review)
Time Frame: 180 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants | 10 | 19

7. Primary Outcome: Frequency of Positive Urine Tests Within 30 Days (Self-report)
Description: Frequency of positive urine tests within 30 days after intervention (data obtained via self-report)
Time Frame: 30 days post intervention
Population: Patient self-report data was not collected due to logistical challenges including COVID-19.
Groups:
- Team Intervention Arm: Recovery coaches and trained health educators will team together and meet with participants (remotely/electronically and/or by phone or in person, when appropriate) at least twice and for a maximum of 7 times. This includes access to mediation, trained mental healthcare providers, and educational resources.
  Team Intervention: The Team will meet with participants (remotely/electronically and/or by phone) and will ask that they select one of three options that may help with opioid addiction:
  1. treatment with buprenorphine/naloxone (BUP),
  2. inpatient, 12-step, or methadone regimens, or
  3. education only (materials provided by the CT Community for Addiction Recovery (CCAR)).
  Throughout the study, participants may switch to any other option.
Arm/Group | Team Intervention Arm
Number analyzed (Participants) | 0

8. Primary Outcome: Frequency of Positive Urine Tests Within 180 Days (Self-report)
Description: Frequency of positive urine tests within 180 days after intervention (data obtained via self-report)
Time Frame: 180 days post intervention
Population: Patient self-report data was not collected due to logistical challenges including COVID-19.
Arm/Group | Team Intervention Arm
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Positive Urine Tests at 30 Days (Chart Review)
Description: Percentage of patients with at least 1 positive urine test at 30 days after intervention (data obtained via chart review)
Time Frame: 30 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants | 1 | 0

10. Secondary Outcome: Percentage of Positive Urine Tests at 180 Days (Chart Review)
Description: Percentage of patients with at least 1 positive urine test at 180 days after intervention (data obtained via chart review)
Time Frame: 180 days post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
Number analyzed (Participants) | 36 | 45
Participants | 5 | 3

11. Secondary Outcome: Percentage of Positive Urine Tests Within 30 Days (Self-report)
Description: Percentage of positive urine tests within 30 days after intervention (data obtained via chart review)
Time Frame: 30 days post intervention
Population: Patient self-report data was not collected due to logistical challenges including COVID-19.
Arm/Group | Team Intervention Arm
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Positive Urine Tests Within 180 Days (Self-report)
Description: Percentage of positive urine tests within 180 days after intervention (data obtained via self-report)
Time Frame: 180 days post intervention
Population: Patient self-report data was not collected due to logistical challenges including COVID-19.
Arm/Group | Team Intervention Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 180 Days
Description: All cause mortality was the only adverse event collected using chart review. Serious and Other [Not Including Serious] Adverse Events were not collected.
Arm/Group | SafetyNet Without Successful Follow Ups | SafetyNet With Successful Follow Ups
All-Cause Mortality (participants affected / at risk) | 2/36 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04253782/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT04253782/ICF_001.pdf